CLINICAL TRIAL: NCT04634253
Title: A Phase 2 Study to Evaluate the Efficacy and Safety of LY3462817 in Participants With Moderately to Severely Active Rheumatoid Arthritis
Brief Title: A Study of LY3462817 in Participants With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17424; J1A-MC-KDAD (Other: Eli Lilly and Company); 2020-002673-10 (EudraCT Number)
Record Dates: First submitted 2020-11-17; First posted 2020-11-18 (Actual); Results first posted 2023-02-01 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-06-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY3462817 300 mg (Experimental): Participants received Intravenous (IV) infusion of 300 mg LY3462817 solution.
  Interventions: Drug: LY3462817
- LY3462817 700 mg (Experimental): Participants received IV infusion of 700 mg LY3462817 solution.
  Interventions: Drug: LY3462817
- Placebo (Placebo Comparator): Participants received IV infusion of 0.9% sodium chloride solution (Placebo).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Given IV
  Arms: Placebo
Drug: LY3462817 — Given IV
  Arms: LY3462817 300 mg; LY3462817 700 mg

SUMMARY:
The reason for this study is to see if the study drug LY3462817 is safe and effective in participants with moderately to severely active rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of adult onset RA as defined by the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria for at least 3 months prior to screening
* Have moderately to severely active RA defined by the presence of ≥6 swollen joints (based on 66 joint count) and ≥6 tender joints (based on 68 joint count) at screening and baseline. The distal interphalangeal joint should be evaluated but not included in the total count to determine eligibility
* Have at least 1 of the following:

  * positive test results for rheumatoid factor or anti-citrullinated peptide antibodies at screening, OR
  * previous radiographs documenting bony erosions in hands or feet consistent with RA
* Have C-reactive protein (CRP) >1.2 times upper limit of normal (ULN) per the central laboratory at screening
* Demonstrated an inadequate response to, or loss of response or intolerance to:

  * at least 1 conventional synthetic disease-modifying antirheumatic drug (csDMARD) treatment OR
  * at least 1 biologic DMARD/tsDMARD treatment

Exclusion Criteria:

* Class IV RA according to ACR revised response criteria
* Have a diagnosis or history of malignant disease within 5 years prior to baseline, with the exceptions of:

  * basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years, or
  * cervical carcinoma in situ, with no evidence of recurrence within the 5 years prior to baseline
* Have presence of confirmed cervical dysplasia
* Have had various types of infection within 3 months of screening or develops any of these infections before the randomization visit.
* Have any of the following:

  * Human immunodeficiency virus (HIV) infection
  * Current infection with hepatitis B virus (HBV) (i.e., positive for hepatitis B surface antigen and/or polymerase chain reaction (PCR) positive for HBV DNA
  * Current infection with hepatitis C virus (HCV) (i.e., positive for HCV RNA)
  * Active tuberculosis (TB)
* Have failed more than 2 biologic DMARDs (bDMARDs) or tsDMARDs (e.g. excluded if have received 2 bDMARDs and 1 tsDMARD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (26):
- United States (7):
  - Arizona Arthritis & Rheumatology Associates, P. C., Mesa, Arizona
  - Arizona Arthritis & Rheumatology Associates, P. C., Phoenix, Arizona
  - Desert Medical Advances, Palm Desert, California
  - Inland Rheumatology & Osteoporosis Medical Group, Upland, California
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
- Czechia (2):
  - Medical Plus, Uherské Hradiště, Zlín
  - PV Medical Services s.r.o., Zlín
- Hungary (5):
  - CRU Hungary Kft., Miskolc, Borsod-Abauj Zemplen county
  - Revita Clinic, Budapest, Pest County
  - Vital Medical Center, Veszprém, Veszprém City
  - Budai Irgalmasrendi Korhaz, Budapest
  - Clinexpert Egeszsegugyi Szolgaltato es Kereskedelmi Kft., Budapest
- Mexico (5):
  - Centro Medico del Angel, Mexicali, Estado de Baja California
  - Centro de Estudios de Investigacion Basica y Clinica, S.C., Guadalajara, Jalisco
  - RM Pharma Specialists S.A. de C.V., Mexico City, Mexico City
  - Köhler & Milstein Research, Mérida, Yucatán
  - Investigacion y Biomedicina de Chihuahua, Chihuahua City
- Poland (4):
  - Klinika Reumatologii i Ukladowych Chorob Tkanki Lacznej, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Twoja Przychodnia Centrum Medyczne Nowa Sol, Nowa Sól, Lubusz Voivodeship
  - Reumatika - Centrum Reumatologii, Warsaw, Masovian Voivodeship
  - Nzoz Bif-Med, Bytom, Silesian Voivodeship
- Puerto Rico (2):
  - Centro Reumatologico Caguas, Caguas
  - Latin Clinical Trial Center, San Juan
- Royal Free Hospital, Barnet, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting
Access Criteria: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting
URL: http://vivli.org/

REFERENCES:
- [Derived] Tuttle J, Emery P, Nirula A. Phase 2 Trial of Peresolimab for Adults with Rheumatoid Arthritis. Reply. N Engl J Med. 2023 Jul 27;389(4):378-379. doi: 10.1056/NEJMc2307020. No abstract available. PMID 37494493
- [Derived] Tuttle J, Drescher E, Simon-Campos JA, Emery P, Greenwald M, Kivitz A, Rha H, Yachi P, Kiley C, Nirula A. A Phase 2 Trial of Peresolimab for Adults with Rheumatoid Arthritis. N Engl J Med. 2023 May 18;388(20):1853-1862. doi: 10.1056/NEJMoa2209856. PMID 37195941
- See also: A Study of LY3462817 in Participants With Rheumatoid Arthritis — https://trials.lillytrialguide.com/en-US/trial/5XEBVhZJQJiPOegLRVANvY

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a Phase 2, proof-of-concept, placebo-controlled, double-blind, randomized study. Participants were randomized to receive LY3462817 700 mg, LY3462817 300 mg, or placebo in an allocation ratio of 2:1:1.
Groups:
- Placebo: Participants received intravenous (IV) infusion of 0.9% sodium chloride solution (Placebo).
- LY3462817 300 mg: Participants received IV infusion of 300 milligrams (mg) LY3462817 solution.
Period: Overall Study
Arm/Group | Placebo | LY3462817 300 mg | LY3462817 700 mg
Started | 24 | 25 | 49
Received at Least One Dose | 24 | 25 | 49
Completed | 22 | 23 | 46
Not Completed | 2 | 2 | 3
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- LY3462817 300 mg: Participants received IV infusion of 300 mg LY3462817 solution.
- Total: Total of all reporting groups
Arm/Group | Placebo | LY3462817 300 mg | LY3462817 700 mg | Total
Number analyzed (Participants) | 24 | 25 | 49 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (11.1) | 50.1 (15.8) | 50.5 (11.2) | 51.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 43 | 82
  Male | 5 | 5 | 6 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 10 | 13 | 30
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 17 | 15 | 34 | 66
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 8 | 5 | 15 | 28
  United States | 4 | 5 | 9 | 18
  Czechia | 0 | 3 | 1 | 4
  Poland | 5 | 2 | 11 | 18
  Mexico | 7 | 10 | 13 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on the Disease Activity Score Modified to Include the 28 Diarthrodial Joint Count-High-Sensitivity C-Reactive Protein (DAS28-hsCRP)
Description: Disease Activity Score (DAS) based on a 28 joint count hsCRP consisted of composite numerical score of the following variables: tender joint count (TJC28), swollen joint count (SJC28), hsCRP (mg/mL), and participant's global assessment of disease activity. DAS28-hsCRP was calculated using following formula: DAS28-hsCRP equals to (=) 0.56*square root (sqrt) (TJC28) plus (+) 0.28*sqrt (SJC28)+ 0.014* participant's global assessment of disease activity + 0.36*natural log(hsCRP+1) +0.96. Scores ranged 1.0-9.4, where lower scores indicated less disease activity. Least Square Mean (LS Mean) was calculated using mixed model repeated measures (MMRM) with treatment, strata (previous RA therapy population), baseline value, visit, treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose and had data for DAS28-hsCRP
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | LY3462817 300 mg | LY3462817 700 mg
Number analyzed (Participants) | 20 | 22 | 42
Units on a scale | -0.99 (0.261) | -1.88 (0.249) | -2.09 (0.184)
Statistical Analysis 1: Comparison: Placebo vs LY3462817 300 mg; Test type: Superiority; p = 0.017, Mixed Models Analysis; LS Mean = -0.88, 95% CI 2-sided [-1.60 to -0.16], Standard Error of Mean 0.361
Statistical Analysis 2: Comparison: Placebo vs LY3462817 700 mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean = -1.09, 95% CI 2-sided [-1.73 to -0.46], Standard Error of Mean 0.320

2. Secondary Outcome: Percentage of Participants Achieving 20% Improvement in American College of Rheumatology Criteria (ACR20)
Description: ACR responders are participants with at least 20% improvement from baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: Health Assessment Questionnaire-Disability Index (HAQ-DI) which measures participants perceived degree of difficulty performing daily activities, acute phase reactant as measured by hsCRP, Patient's Assessment of Pain-Visual Analog Scale (Pain-VAS), Patient's Global Assessment of Disease Activity (PaGADA_VAS), and Physician's Global Assessment of Disease Activity (PhGADA_VAS).
Time Frame: Week 12
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | LY3462817 300 mg | LY3462817 700 mg
Number analyzed (Participants) | 24 | 25 | 49
Percentage of Participants | 41.7 [21.9 to 61.4] | 44.0 [24.5 to 63.5] | 71.4 [58.8 to 84.1]
Statistical Analysis 1: Comparison: Placebo vs LY3462817 300 mg; Test type: Superiority; p = 0.997, Regression, Logistic; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.29 to 3.44]
Statistical Analysis 2: Comparison: Placebo vs LY3462817 700 mg; Test type: Superiority; p = 0.032, Regression, Logistic; Odds Ratio (OR) = 3.40, 95% CI 2-sided [1.11 to 10.40]

3. Secondary Outcome: Percentage of Participants Achieving 70% Improvement in American College of Rheumatology Criteria (ACR70)
Description: ACR responders are participants with at least 70% improvement from baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: Health Assessment Questionnaire-Disability Index (HAQ-DI) which measures participants perceived degree of difficulty performing daily activities, acute phase reactant as measured by hsCRP, Patient's Assessment of Pain-Visual Analog Scale (Pain-VAS), Patient's Global Assessment of Disease Activity (PaGADA_VAS), and Physician's Global Assessment of Disease Activity (PhGADA_VAS).
Time Frame: Week 12
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | LY3462817 300 mg | LY3462817 700 mg
Number analyzed (Participants) | 24 | 25 | 49
Percentage of Participants | 16.7 [1.8 to 31.6] | 4.0 [0 to 11.7] | 20.4 [9.1 to 31.7]
Statistical Analysis 1: Comparison: Placebo vs LY3462817 300 mg; Test type: Superiority; p = 0.235, Regression, Logistic; Odds Ratio (OR) = 0.29, 95% CI 2-sided [0.04 to 2.25]
Statistical Analysis 2: Comparison: Placebo vs LY3462817 700 mg; Test type: Superiority; p = 0.661, Regression, Logistic; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.33 to 5.61]

4. Secondary Outcome: Percentage of Participants Achieving 50% Improvement in American College of Rheumatology Criteria (ACR50)
Description: ACR responders are participants with at least 50% improvement from baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: Health Assessment Questionnaire-Disability Index (HAQ-DI) which measures participants perceived degree of difficulty performing daily activities, acute phase reactant as measured by hsCRP, Patient's Assessment of Pain-Visual Analog Scale (Pain-VAS), Patient's Global Assessment of Disease Activity (PaGADA_VAS), and Physician's Global Assessment of Disease Activity (PhGADA_VAS).
Time Frame: Week 12
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | LY3462817 300 mg | LY3462817 700 mg
Number analyzed (Participants) | 24 | 25 | 49
Percentage of Participants | 20.8 [4.6 to 37.1] | 20.0 [4.3 to 35.7] | 38.8 [25.1 to 52.4]
Statistical Analysis 1: Comparison: Placebo vs LY3462817 300 mg; Test type: Superiority; p = 0.965, Regression, Logistic; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.22 to 4.28]
Statistical Analysis 2: Comparison: Placebo vs LY3462817 700 mg; Test type: Superiority; p = 0.098, Regression, Logistic; Odds Ratio (OR) = 2.91, 95% CI 2-sided [0.82 to 10.33]

5. Secondary Outcome: Change From Baseline for Mean Simplified Disease Activity Index (SDAI)
Description: The SDAI is a tool for measurement of disease activity in RA that integrates measures of physical examination, acute phase response, patient self-assessment, and evaluator assessment. The SDAI is calculated by adding together scores from 1) TJC28 (0 to 28), 2) SJC28 (0 to 28), 3) acute phase response using C-reactive protein (0.1 to 10.0 mg/dL), 4) Patient's Global Assessment of Disease Activity using VAS (0 to 10 cm), and 5) Physician's Global Assessment of Disease Activity using VAS (0 to 10 cm). Total Score scale range is 0 (remission) to 86 (high disease activity). LS Mean was calculated using mixed model repeated measures (MMRM) with treatment, strata (previous RA therapy population), baseline value, visit, treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose and had data for SDAI.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY3462817 300 mg | LY3462817 700 mg
Number analyzed (Participants) | 20 | 21 | 42
units on a scale | -13.80 (2.664) | -25.06 (2.571) | -26.90 (1.880)
Statistical Analysis 1: Comparison: Placebo vs LY3462817 300 mg; Test type: Superiority; p = 0.003, Mixed Models Analysis; LS Mean Difference = -11.26, 95% CI 2-sided [-18.65 to -3.87], Standard Error of Mean 3.710
Statistical Analysis 2: Comparison: Placebo vs LY3462817 700 mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -13.10, 95% CI 2-sided [-19.61 to -6.60], Standard Error of Mean 3.265

6. Secondary Outcome: Change From Baseline for Mean Clinical Disease Activity Index (CDAI)
Description: The CDAI is a tool for measurement of disease activity in RA that does not require a laboratory component and was scored by the investigative site. It integrates TJC28 (scored 0-28 with higher scores indicating higher disease activity), SJC28 (scored 0-28 with higher scores indicating higher disease activity), Patient's Global Assessment of Disease Activity (scored on a visual analogue scale from 0-10 cm with higher scores indicating higher disease activity), and Physician's Global Assessment of Disease Activity (scored on a visual analogue scale from 0-10 cm with higher scores indicating higher disease activity). The CDAI is calculated by summing the values of the 4 components. CDAI scores range from 0 to 76; lower scores indicated lower disease activity. A negative change from baseline indicates improvement in condition. LS Mean was calculated using MMRM with treatment, strata (previous RA therapy population), baseline value, visit, treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose and had data for CDAI.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY3462817 300 mg | LY3462817 700 mg
Number analyzed (Participants) | 20 | 21 | 44
units on a scale | -13.75 (2.709) | -24.06 (2.628) | -25.51 (1.854)
Statistical Analysis 1: Comparison: Placebo vs LY3462817 300 mg; Test type: Superiority; p = 0.008, Mixed Models Analysis; LS Mean Difference = -10.30, 95% CI 2-sided [-17.83 to -2.77], Standard Error of Mean 3.782
Statistical Analysis 2: Comparison: Placebo vs LY3462817 700 mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -11.76, 95% CI 2-sided [-18.29 to -5.22], Standard Error of Mean 3.282

7. Secondary Outcome: Change From Baseline in Mental Component Score (MCS), Physical Component Score (PCS) of the Medical Outcomes Study 36-Item Short Form Health Survey Version 2 Acute (SF-36v2 Acute)
Description: The SF-36 is a health-related survey that assesses participant's health status and consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems, role limitations due to emotional problems, general health, mental health, social functioning, and vitality. The 8 domains are combined to form 2 component scores mental (MCS) and physical (PCS). MCS consisted of social functioning, vitality, mental health, and role-emotional scales. PCS consisted of physical functioning, bodily pain, role-physical, and general health scales. Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale with higher scores indicating better health status. LS mean was determined by ANCOVA with factors for treatment and previous RA therapy population included as fixed factors,
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose and had data for MCS and PCS.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | LY3462817 300 mg | LY3462817 700 mg
Number analyzed (Participants) | 21 | 23 | 47
Units on a scale
  MCS | 3.48 (1.715) | 0.55 (1.630) | 4.64 (1.166)
  PCS | 5.01 (1.711) | 7.03 (1.633) | 6.43 (1.165)
Statistical Analysis 1: Comparison: Placebo vs LY3462817 300 mg; Mental Component Score (MCS); Test type: Superiority; p = 0.218, ANCOVA; LS Mean Difference = -2.93, 95% CI 2-sided [-7.63 to 1.77], Standard Error of Mean 2.365
Statistical Analysis 2: Comparison: Placebo vs LY3462817 700 mg; Mental Component Score (MCS); Test type: Superiority; p = 0.578, ANCOVA; LS Mean Difference = 1.15, 95% CI 2-sided [-2.95 to 5.26], Standard Error of Mean 2.065
Statistical Analysis 3: Comparison: Placebo vs LY3462817 300 mg; Physical Component Score (PCS); Test type: Superiority; p = 0.396, ANCOVA; LS Mean Difference = 2.02, 95% CI 2-sided [-2.69 to 6.73], Standard Error of Mean 2.368
Statistical Analysis 4: Comparison: Placebo vs LY3462817 700 mg; Physical Component Score (PCS); Test type: Superiority; p = 0.493, ANCOVA; LS Mean Difference = 1.42, 95% CI 2-sided [-2.67 to 5.50], Standard Error of Mean 2.057

8. Secondary Outcome: Pharmacokinetics (PK): Observed Concentration of LY3462817
Description: PK: Observed Concentration of LY3462817
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Median (95% Confidence Interval); unit: nanograms per milliliter
Arm/Group | LY3462817 300 mg | LY3462817 700 mg
Number analyzed (Participants) | 25 | 49
nanograms per milliliter | 7970 [1290 to 17100] | 15600 [1820 to 36600]

ADVERSE EVENTS:
Time Frame: Baseline, up to Week 12
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Placebo | LY3462817 300 mg | LY3462817 700 mg
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25 | 1/49
Other Adverse Events (participants affected / at risk) | 9/24 | 8/25 | 13/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | LY3462817 300 mg (N=25) | LY3462817 700 mg (N=49)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=24) | LY3462817 300 mg (N=25) | LY3462817 700 mg (N=49)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0/19 (0) | 0/20 (0) | 1/43 (1)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Allodynia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (3)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
No adjustment for multiplicity was made. For assessments beyond the primary endpoint, nominal p-values are reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT04634253/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/53/NCT04634253/SAP_001.pdf